CLINICAL TRIAL: NCT01151085
Title: Vfend Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Voriconazole (Vfend) Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501076
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-05

CONDITIONS: Systemic Mycosis
Keywords: Systemic Mycosis; Aspergillus infection; Candidiasis; Cryptococcal infections; Japanese; voriconazole; VFEND; Regulatory Post Marketing Commitment Plan.
MeSH Terms: conditions — Aspergillosis; Candidiasis | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Voriconazole: Subjects who are treated with voriconazole
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Voriconazole Intravenous Solution 200 mg:
  Voriconazole is administered by intravenous drip infusion at the dose of 6 mg/kg twice daily on day 1 and 3 mg/kg or 4 mg/kg twice daily from day 2 onward in adults.
  Voriconazole Tablet 50 mg/ Voriconazole Tablet 200 mg:
  administration for an adult (weighing 40 kg or more) is voriconazole 300mg orally twice daily between meals for day 1 and then 150 mg or 200 mg twice daily between meals from day 2 onward.
  Depending on the symptoms or in cases where the effect is insufficient, the dosage may be increased.
  However, the maximum dose on day 1 must be 400 mg twice daily, and the maximum dose from day 2 onward must be 300 mg twice daily.
  In patients weighing less than 40 kg, voriconazole 150 mg shall be administered twice daily on day 1, and voriconazole 100 mg shall be administered twice daily from day 2 onward.
  Depending on the symptoms, the maintenance dose from day 2 onward may be increased to 150 mg twice daily.
  Other Names: VFEND for Intravenous Use, Voriconazole for Intravenous Use, VFEND Tablets, Voriconazole Tablet

SUMMARY:
To collect the efficacy and safety informations of voriconazole related to their appropriate use in daily practice.

DETAILED DESCRIPTION:
All the subjects whom an investigator prescribes the first voriconazole (VFEND) should be registered consecutively until the number of subjects reaches target number in order to extract subjects enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects intend to treat their deep mycosis who are prescribed voriconazole (VFEND) by their Physicians.

Exclusion Criteria:

* Subject who heve been prescribed voriconazole (VFEND) before.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A1501076 prescribes the voriconazole (VFEND).
Sampling Method: Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2006-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501076&StudyName=Voriconazole%20%28Vfend%29%20Drug%20Use%20Investigation%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Voriconazole: Participants taking Voriconazole according to Japanese Package Insert.
Period: Overall Study
Arm/Group | Voriconazole
Started | 1002
Completed | 946
Not Completed | 56
Not completed — Lost to Follow-up | 31
Not completed — Protocol Violation | 25

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole
Number analyzed (Participants) | 946
Age, Customized [Number; unit: participants]
  <65 years | 500
  >=65 years | 446
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335
  Male | 611

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Frequency of Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Voriconazole, irrespective of causal relationship to Voriconazole (including clinically problematic abnormal changes in laboratory test values). Treatment related Adverse Events were evaluated in company with the causal relationship to Voriconazole.
Time Frame: 16 weeks
Population: No statistical analysis provided for the frequency of treatment related adverse events.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 946
participants | 220

2. Primary Outcome: Number of Participants That Responded to Voriconazole Treatment.
Description: The primary endpoint was the efficacy ratio (number of effective cases/number of evaluable cases for efficacy assessment) among the cohort comprising the subjects for efficacy analysis.
Time Frame: 16 weeks
Population: The efficacy analysis population basically consists of the evaluable cases in accordance with the separately prepared analysis plan (cases judged to have been evaluated appropriately).
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 558
participants | 405

3. Secondary Outcome: Number of Unlisted Treatment Related Adverse Events in Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in participants after administration of Voriconazole, irrespective of causal relationship to Voriconazole (including clinically problematic abnormal changes in laboratory test values). Number of Treatment Related Adverse Events were evaluated in company with the causal relationship to Voriconazole. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: 16 weeks
Population: No statistical analysis provided for the number of the unlisted treatment related adverse events in Japanese Package Insert.
Measure: Number; unit: events
Arm/Group | Voriconazole
Number analyzed (Participants) | 946
events | 19

4. Secondary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Gender.
Description: Number of participants with Treatment Related Adverse Events of Voriconazole to determine whether male or female is significant risk factor.
Time Frame: 16 weeks
Population: The safety analysis population consists of the cases that satisfy the cases conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Groups:
- Male: Male Participants taking Voriconazole according to Japanese Package Insert.
- Female: Female Participants taking Voriconazole according to Japanese Package Insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 611 | 335
participants | 156 | 64
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is there is no difference between "Male and Female " in the Frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p = 0.030, Fisher Exact

5. Secondary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Severity of Infections.
Description: Number of participants with Treatment Related Adverse Events of Voriconazole to determine whether severity of infections(mild, moderate or severe) is significant risk factor.
Time Frame: 16 weeks
Measure: Number; unit: participants
Groups:
- Mild Infection: Participants with mild infection who taking Voriconazole according to Japanese Package Insert.
- Moderate Infection: Participants with moderate infection who taking Voriconazole according to Japanese Package Insert.
- Severe Infection: Participants with severe infection who taking Voriconazole according to Japanese Package Insert.
Arm/Group | Mild Infection | Moderate Infection | Severe Infection
Number analyzed (Participants) | 229 | 412 | 305
participants | 60 | 115 | 45
Statistical Analysis 1: Comparison: Mild Infection vs Moderate Infection vs Severe Infection; The risk factor tested was "Severity of infections". The null hypothesis is there is no difference among "mild, moderate and severe" in the Frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Secondary Outcome: Risk Factors for the Frequency of Treatment Related Adverse Events -Past History.
Description: Number of participants with Treatment Related Adverse Events of Voriconazole to determine whether with or without Past History is significant risk factor.
Time Frame: 16 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- With Past History: Participants with Past History who taking Voriconazole according to Japanese Package Insert.
- Without Past History: Participants without Past History who taking Voriconazole according to Japanese Package Insert.
Arm/Group | With Past History | Without Past History
Number analyzed (Participants) | 271 | 673
participants | 77 | 142
Statistical Analysis 1: Comparison: With Past History vs Without Past History; The risk factor tested was "Past History". The null hypothesis is there is no difference between "with and without Past History" in the Frequency of Treatment Related Adverse Events; Test type: Superiority or Other; p = 0.017, Fisher Exact

7. Secondary Outcome: Number of Participants That Responded to Voriconazole Treatment -Severity of Infections.
Description: Number of participants that responded to voriconazole to determine whether severity of infections(mild, moderate or severe) is significant risk factor.
Time Frame: 16 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Mild Infection | Moderate Infection | Severe Infection
Number analyzed (Participants) | 129 | 269 | 160
participants | 106 | 202 | 97
Statistical Analysis 1: Comparison: Mild Infection vs Moderate Infection vs Severe Infection; Statistical Analysis for Risk Factors for the Proportion of Responders to Voriconazole treatment -Severity of infections; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events during the study.
Arm/Group | Voriconazole
Serious Adverse Events (participants affected / at risk) | 24/946
Other Adverse Events (participants affected / at risk) | 201/946
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voriconazole (N=946)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4)
Liver disorder (Hepatobiliary disorders) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Drug interaction (General disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voriconazole (N=946)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 11 (11)
Hallucination, visual (Psychiatric disorders) | 3 (3)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Eyelid disorder (Eye disorders) | 1 (1)
Colour blindness acquired (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 9 (9)
Chromatopsia (Eye disorders) | 3 (3)
Vision blurred (Eye disorders) | 6 (6)
Photophobia (Eye disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 57 (57)
Liver disorder (Hepatobiliary disorders) | 26 (26)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3)
Renal disorder (Renal and urinary disorders) | 2 (2)
Colour blindness (Congenital, familial and genetic disorders) | 2 (2)
Feeling abnormal (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Alanine aminotransferase increased (Investigations) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 16 (16)
Liver function test abnormal (Investigations) | 5 (5)
Hepatic enzyme increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 11 (11)
Blood creatinine increased (Investigations) | 3 (3)
Blood creatine increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (3)
Blood urea increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.